CLINICAL TRIAL: NCT02999165
Title: Breastfeeding Infants Receiving Respiratory Support Trial
Acronym: BIRRST
Status: Terminated | Type: Observational
Why Stopped: Failure to recruit participants due to change in local clinical practice.
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 16/WS/0142
Record Dates: First submitted 2016-11-01; First posted 2016-12-21 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Intensive Care, Neonatal; Neonatal Respiratory Distress Syndrome; Continuous Positive Airway Pressure; Breast Feeding; Infant, Premature
Keywords: Breastfeeding; CPAP; Humidified High Flow Nasal Cannula Oxygen; preterm neonate
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Breast Feeding; Premature Birth | interventions — Lactation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CPAP group: 25 infants undergoing treatment with continuous nCPAP who are making attempts at breast feeding and receiving nasogastric feeds.
  Interventions: Other: Breast feeding; Other: Nasogastric feeding
- HHFNC group: 25 infants undergoing treatment with continuous HHFNC oxygen who are making attempts at breast feeding and receiving nasogastric feeds.
  Interventions: Other: Breast feeding; Other: Nasogastric feeding

INTERVENTIONS:
Other: Breast feeding — Infants on respiratory support will be allowed to attempt to breast feed (with a top up nasogastric tube feed if required).
Other: Nasogastric feeding — The control intervention is feeding via nasogastric tube

SUMMARY:
The purpose of this study is to assess whether two methods of breathing support in babies called 'Humidified High-Flow Nasal Cannula' oxygen (HHFNC) and 'nasal Continuous Positive Airways Pressure' (nCPAP) are compatible with breastfeeding. Many babies who are premature or unwell after birth require help with their breathing. This is often achieved by blowing a continuous flow of air through the nose and down into the lungs in order to reduce the amount of effort the baby needs to inflate the lungs during breathing.

Currently some centres allow babies to breastfeed whilst undergoing breathing support whilst other centres do not in case there is an increased risk of choking or other harmful events. In the latter case, babies are fed using a nasogastric tube (NGT) that runs from the baby's nostrils into their stomach.

At this centre, babies are allowed to breastfeed whilst simultaneously on either HHFNC or nCPAP. This is because the concerns over the choking risk are not evidence based. This study aims to conclusively prove that thisfeeding protocol is safe and then to expand into other areas of research to find out the following:

* Whether breastfeeding during nCPAP or HHFNC leads to babies establishing full breastfeeding sooner (and subsequently reduce the length of their stay in hospital)
* What the effects of breastfeeding of nCPAP or HHFNC are on a baby's parents (e.g. whether it enhances bonding)
* If nCPAP and HHFNC have different effects on breastfeeding As part of this study the investigators will observe stable babies on nCPAP or HHFNC during breastfeeding episodes. The investigators will monitor the babies for signs of distress or instability and whether they are more stable when breastfeeding is not occurring. This will be compared to an episode where the same baby is fed by NGT to see which technique is better.

DETAILED DESCRIPTION:
BACKGROUND Breastfeeding infants receiving respiratory support (nCPAP or HHFNC) is a controversial topic. Expert consensus has been that feeding should be delayed until respiratory support (including nCPAP or HHFNC) is no longer needed. Data from animal models suggests that nasal CPAP can affect swallowing behaviour in infant animals but the magnitude and clinical significance of any effect is unclear even in animals. Studies in adults are also lacking but some have shown that swallowing can be impaired during CPAP therapy. There is no research into whether HHFNC has similar effects in any of the above populations. There is currently no published data on the safety or efficacy of breastfeeding infants receiving respiratory support via nasal CPAP or HHFNC.

nCPAP is a key intervention in the current care of many babies as it is the preferred mode of non-invasive respiratory support and compared to conventional mechanical ventilation it has been shown to reduce the incidence of bronchopulmonary dysplasia . HHFNC oxygen has emerged as another method of respiratory support. It has been shown that it is non-inferior to nCPAP following extubation although it is clear that the mechanics of flow delivery differ from nCPAP. There is some evidence that HHFNC use is associated with a reduction in some adverse effects when compared with nCPAP, such as nasal trauma.

Some infants, especially infants born very preterm, spend prolonged periods on nasal CPAP or HHFNC. Normal oral feeding is often delayed in these children because respiratory support is needed. It has been shown that premature infants can show breastfeeding cues from a very early stage and if infants are given the opportunity breastfeeding can be well established. Recent studies have shown that early introduction of oral feeding in preterm neonates is not associated with adverse outcomes and leads to earlier establishment of full oral feeding and discharge home.

RATIONALE FOR CURRENT STUDY There is uncertainty surrounding the safety of breastfeeding babies on nasal nCPAP or HHFNC. There is great disparity in clinical practice between neonatal units. At our department babies on respiratory support have traditionally been offered the chance to breastfeed. Local experience is that this is not associated with adverse events. When compared to other units internationally (as part of the Vermont-Oxford Network of neonatal units) our unit does not have an excess of complications due to this practice.

Establishing the safety of breastfeeding whilst receiving nCPAP or HHFNC will provide clinicians with the information necessary to decide when breastfeeding should be attempted in infants needing ongoing respiratory support.

In addition the study team want to use this opportunity to establish the feasibility of future studies. If breastfeeding on nCPAP and HHFNC is safe the study team want to prepare for further investigation in this field looking at:

* Whether infants being breastfed on nCPAP and HHFNC can show progression from immature to mature feeding behaviours and if this ultimately leads to earlier establishment of full oral feeding.
* What impact being breastfed on nCPAP or HHFNC has on the parents of these babies. If breastfeeding on nCPAP and HHFNC help bonding this would be another important factor to consider.
* To prepare to compare HHFNC and nCPAP to see if the effects they have on breastfeeding differ. If nCPAP or HHFNC is superior to the other this may affect clinician decision on which to use.

Clarity in this field will enable clinicians to make safe decisions about when infants receiving respiratory support should be allowed to breastfeed aiding delivery of optimal care.

STUDY OBJECTIVES The primary objective of this prospective observational study is to test the hypothesis that breastfeeding infants undergoing nCPAP or HHFNC is safe.

The secondary objective is to test the feasibility of future studies:

* To investigate the feasibility of testing the hypothesis that breastfeeding preterm infants while treated with nCPAP or HHFNC leads to faster establishment of full enteral feeds as this could allow patients to benefit from earlier discharge home. This study will show whether the methods used are acceptable to parents and capture the outcome data required. Data gathered will give information on the standard deviation of outcomes to enable accurate sample size calculation.
* To investigate the feasibility of assessing parental perception of breastfeeding babies receiving respiratory support and the effect it has on bonding. Questionnaire responses and feedback from parents will be reviewed to investigate their feeidng issues and concerns.
* To investigate the feasibility of comparing nCPAP and HHFNC to evaluate whether they have different effects breastfeeding for infants.

STUDY DESIGN Prospective, observational, single centre safety study. Recruitment will occur over a one-year period. Parents will initially be approached by members of the healthcare team. With their consent they will then be contacted by a member of the BIRRST team and informed about the details of the study. Written consent from the parents must be obtained in order to include a patient. It will be explained to parents that it is common practise to offer infants to be breast fed while still on respiratory support in this unit.

No change will be made to the management of babies enrolled in this study. Babies will be observed during feeding episodes but the timing of these feeds, whether a baby will be fed by breastfeeding or NGT and all details relating to how a feed is administered are decisions that will be made by the nursing team looking after a baby (in conjunction with the baby's parents). The study team will have no influence or say in these decisions and will just observe standard practice for this unit.

50 infants will be recruited, 25 infants treated with nCPAP and 25 infants treated with HHFNC while breast feeding attempts are made. Each child is estimated to have between 4 and 6 observations. There will be no crossover between the respiratory support modalities. Infants without any respiratory support will no longer be eligible or included in the study.

130 paired observations of breastfeeding and NGT feeding during nCPAP treatment will be made. In addition 130 paired observations of breastfeeding and NGT feeding while babies are on HHFNC will be made. Each infant will serve as its own control as feeding episodes will be paired so that a breastfeed and an NGT feed are both observed within a 12 hour period. This will minimise variation caused by changes in the infants' condition.

It is unlikely that infants will be able to obtain sufficient volume of milk while learning to breastfeed and so after each breastfeeding attempt the babies will be offered a top-up via NGT to ensure they receive their required feed volume.

Once a baby is enrolled in the study feeding episodes will be regularly observed (as is feasible with respect to staff availability and parental presence). If a baby is too unwell to be observed this will be documented.

Prior to the observation the baby's stability during the preceding hour will be evaluated and recorded. During a feeding episode all infants will be directly observed for a 30 minute period during which they will either receive a breast feed with a subsequent NGT top up or solely an NGT feed. Subsequently the baby's stability over the following hour will be retrospectively assessed. All infants will receive continuous nCPAP or HHFNC throughout.

During a feeding episode heart rate and oxygen saturation will be continuously monitored using pulse oximetry. Apnoea monitors will be used to assess episodes of apnoea. Axillary temperature will be assessed at the beginning and end of the feeding episode. The oxygen requirement will be measured from the CPAP/HHFNC machine.

The stability of the neonate during each feeding episode will be compared with their stability over the preceding hour by reviewing the documented incidence of desaturations, bradycardias and apnoeas and the neonate's temperature on their observation chart.

Quality of breastfeeding will be assessed using videos of breastfeeding episodes. These videos will be reviewed by trained assessors (Speech and Language Therapists with an interest in lactation from Imperial College Healthcare NHS Trust) who will use the PIBBS tool to assess the quality of feeding. They will look for feeding behaviours to assess the maturity of feeding.

Serial feeding episodes will be compared to assess whether there is a progression from more immature to mature feeding as the babies have breastfeeding opportunities on CPAP or HHFNC. This data will be used to assess whether future studies in this area to explore how feeding behaviours progress would be beneficial.

It will also be recorded at what corrected gestational age/actual age these babies establish oral feeding; how they are fed at discharge (breast or bottle) and what milk they are discharged home on. This data will allow planning of future studies to assess whether early attempts at breastfeeding whilst receiving CPAP or HHFNC help the establishment of full breastfeeding.

The parental perception of feeding with respiratory support will be assessed using a parental questionnaire. This will use a visual analogue scale to assess whether parents feel that breastfeeding during respiratory support is beneficial to their infants overall care and what impact the feeding opportunities has had on their bonding with their baby. This data will be used to assess the feasibility of further studies in this area by establishing the parental tolerance of breastfeeding babies receiving respiratory support and developing a questionnaire that will effectively explore the parental experience.

The data collected for nCPAP and HHFNC separately will be used to establish the sample size that will be required in future studies to compare the two modalities to see if there are significant differences between the two (in terms of safety, efficacy and parental tolerance).

STATISTICS AND DATA ANALYSIS Analysis of the pilot study data suggested that desaturation was the most common adverse event associated with feeding during nCPAP or HHFNC treatment. The sample size has been calculated to show a significant difference based on the results from the pilot data.

128 feeding episodes are required to get 80% power at the 5% significance level to find a difference in mean duration of desaturation episodes of 1.25 minutes, based on a standard deviation for changes in this outcome of 5 (taken from pilot data). This is felt to be a clinically significant increase in desaturation episodes over a 30 minute period.

The feeding episodes may come from around 25 babies. As each baby acts as its own control (because each breastfeeding episode is paired with an episode of NGT feeding occurring within 24 hours) the sample size is dependent on the number of feeding episodes observed, not the number of babies.

Analysis: paired t-test of mean duration of desaturation. McNemar's test to compared paired proportions between groups.

Data and all appropriate documentation will be stored for 5 years after the completion of the study, including the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Infants cared for at Imperial College Healthcare NHS trust neonatal unit at Queen Charlottes and Chelsea Hospital and St Marys Hospital. Infants will be eligible if they are over 30 weeks of gestational age and receive continuous treatment with nCPAP or HHFNC .

Exclusion Criteria:

* Major congenital malformation or underlying genetic disorder
* signs of severe progressive respiratory distress
* FiO2 > 0.4
* PCo2 > 9kPa
* Need for high CPAP > 8cmH2O
* Need for HHFNC with flow rate of >8litres/min
* Severe temperature instability, not tolerating 30 min outside the incubator
* CPAP or HHFNC treatment stopped

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants requiring medical care on a neonatal unit who are receiving continuous treatment with nCPAP or HHFNC and are making attempts to breast feed
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Incidence of episodes of desaturation during a feeding episode | 30 minutes
  During a feeding episode physiological parameters (heart rate, respiratory rate, oxygen saturation) will be observed continuously using Massimo monitors and recorded every 5 minutes.
  Any episodes of desaturation will be recorded (duration of time that saturations under 92% and lowest recorded saturations).
Incidence of episodes of bradycardia during a feeding episode | 30 minutes
  During a feeding episode physiological parameters (heart rate, respiratory rate, oxygen saturation) will be observed continuously using Massimo monitors and recorded every 5 minutes.
  Any episodes of bradycardia during a feeding episode will be recorded (duration that heart rate is less than 100 beats per minute and lowest recorded heartrate).
Incidence of episodes of apnoea during a feeding episode | 30 minutes
  During a feeding episode physiological parameters (heart rate, respiratory rate, oxygen saturation) will be observed continuously using a Massimo monitor and recorded every 5 minutes.
  Any episodes of apnoea during a feeding episode will be recorded (duration of apnoea).
Incidence of episodes of temperature instability during a feeding episode | 30 minutes
  Temperature will be recorded at beginning and end of a feeding episode (in degrees celsius).
  Any episodes of temperature instability during a feeding episode will be recorded.

SECONDARY OUTCOMES:
Breastfeeding behaviours displayed measured using the PIBBS scale | 30 minutes
  Efficacy of breast feeding will be assessed using the PIBBS scale (Premature Infant Breastfeeding Behaviours Scale)
Parental perception of breast feeding an infant receiving respiratory support | One week
  Parents will complete a questionnaire addressing parental perception of breastfeeding using a series of visual analogue scales.

OTHER OUTCOMES:
Gestational age at full oral feeding | Through study completion, an average of six months
  The age at which each infant achieves full oral feeding will be documented
Route of oral feeding at discharge | Through study completion, an average of six months
  The route of oral feeding (i.e. bottle vs. breast feeding) at the time of discharge home will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rakow, MD, Principal Investigator — Imperial College NHS Trust
Locations (1):
- Queen Charlotte's and Chelsea Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised, non-identifiable data available on request